CLINICAL TRIAL: NCT06422208
Title: A Phase 1 Clinical Trial of Autologous iPSC-Derived Dopamine Neuron Transplantation for Parkinson's Disease
Brief Title: Autologous iPSC-Derived Dopamine Neuron Transplantation for Parkinson's Disease
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Penelope J. Hallett, Ph.D. (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Oryon Cell Therapies (Unknown)
Responsible Party: Sponsor-Investigator, Penelope J. Hallett, Ph.D., Associate Professor, Mclean Hospital
Organization: Mclean Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003609; U01NS109463 (NIH)
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous midbrain dopamine neurons (Experimental)
  Interventions: Biological: Autologous midbrain dopamine neurons

INTERVENTIONS:
Biological: Autologous midbrain dopamine neurons — The autologous midbrain dopamine neurons are a experimental cryopreserved cell product derived from human autologous induced pluripotent stem cells. The autologous midbrain dopamine neurons will be surgically administered into the putamen, unilaterally, in a single surgical session.

SUMMARY:
This research study is evaluating an investigational cell product called autologous induced pluripotent stem cell (iPSC)-derived dopamine neurons. This research study is a single-center Phase 1/2a clinical trial, which will test the safety of injecting the investigational cell product into the brain of subjects with Parkinson's disease.

DETAILED DESCRIPTION:
The goal of this research study is to test a new treatment for Parkinson's disease. Parkinson's disease is a progressive disease that causes people to lose specific brain cells called midbrain dopamine neurons. When these dopamine neurons are lost, it leads to a lack of dopamine in the brain. When there is not enough dopamine, people with Parkinson's disease experience problems with their movement. This trial will test whether new dopamine neurons made from blood cells from subjects with Parkinson's disease are safe when surgically injected into the area of the brain affected (called the putamen) of the same subjects (called autologous transplantation). The trial will assess the safety of the injected cells and will also measure the effects of the transplanted autologous dopamine neurons on Parkinson's disease symptoms.

At this time, autologous iPSC-derived midbrain dopamine neurons are available only through participation in the ongoing Phase 1/2a clinical trial. Expanded access or compassionate use outside of the trial is not available.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages 55 to eighty.
* Diagnosis of Parkinson's disease with motor symptoms by neurologist according to Movement Disorder Society (MDS) 2015 Clinical Diagnostic Criteria for Parkinson's disease.
* Diagnosis of Parkinson's disease for at least 5 years.
* Dopamine drug responsiveness demonstrated by a positive "on/off" test with at least a 30% improvement on UPDRS III (motor) scale.
* No gross abnormalities on MRI, including hydrocephalus or extensive white matter disease.
* No significant cognitive impairment (Montreal Cognitive Assessment).
* No significant untreated depression (Beck Depression Inventory 2).
* Up to date cancer screening per primary MD.
* Able to understand trial requirements and intervention procedures and provide written informed consent.

Exclusion Criteria:

* History of intracranial surgeries.
* Any previous thalamotomy, pallidotomy or deep brain stimulation.
* Atypical Parkinsonism (Parkinsonism-Plus syndrome, secondary parkinsonism, hereditary parkinsonism)
* History of psychiatric disorders including schizophrenia or psychosis likely to compromise with ability to comply with trial protocol requirements.
* Prior history of intracerebral, subdural, or epidural hemorrhage.
* History of malignancy within 5 years.
* Inability to have an MRI.
* Life expectancy < 6 months due to concomitant illnesses.
* Ingestion of investigational drug or recipient of investigational procedure within 6 months prior to trial.
* Subjects with active cardiovascular and cerebrovascular disease within 6 months prior to signing the informed consent form:

  1. History of severe heart failure (congestive heart failure of New York Heart Association Class II or above or left ventricular ejection fraction < 35% by any examination method), unstable angina pectoris and myocardial infarction
  2. Severe arrhythmia
  3. History of cardiovascular surgery (cardiac, vascular stent surgery, angioplasty);
  4. History of stroke or transient ischemic attack
  5. History of subarachnoid hemorrhage
  6. Subjects with major vascular diseases (aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis)
* Hypertensive subjects with poorly controlled blood pressure (defined as blood pressure above 160/100 mmHg despite treatment with antihypertensive drugs) and subjects with severe postural hypotension.
* Abnormal pre-operative coagulation labs.
* Any necessary chronic anticoagulation medication in use (not including antiplatelet therapy and chronic NSAID).
* Diabetic subjects with poorly controlled blood glucose (glycosylated hemoglobin > 9.0%, or fasting plasma glucose (FPG) ≥ 11.1 mmol/L).
* Active infectious disease. Subjects known to have tested positive for HIV, Human T-lymphotropic Virus, Hepatitis B Virus, Hepatitis C Virus, Cytomegalovirus (IgM > IgG) and/or syphilis will be evaluated by an expert as to subject eligibility based on the subject's infectious status.
* Any illness which, in the Investigator's judgment, will interfere with the subject's ability to comply with the protocol, compromise subject safety, or interfere with the interpretation of the trial results.
* Active clinical infection being treated by antibiotics within one week of enrollment.
* Known drug or alcohol dependence or any other clinical factors or conditions (for example, history of seizures) which will interfere with the trial conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Unwilling and/or not able to give written informed consent.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety: number and severity of adverse events and serious adverse events | Baseline to 12 months post-transplant and baseline to 18 months post-transplant
  To assess the safety of autologous transplantation of cryopreserved midbrain dopamine neurons into the putamen of subjects with Parkinson's disease by measuring (1) the incidence of serious adverse events at 12 months and 18 months post-transplantation and (2) the incidence and severity of all intervention emergent adverse events.

SECONDARY OUTCOMES:
Change in UPDRS Part III | 18 months following transplantation
  Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (UPDRS) motor (Part III) compared to the baseline. UPDRS Part III assesses motor function and is measured in both "Off" and "On" states. UPDRS Part III score range: 0-132. A lower score is associated with milder Parkinson's disease motor symptoms.
Change in ON time without troublesome dyskinesia | 18 months following transplantation
  Change in ON time without troublesome dyskinesia is measured using a Parkinson's disease patient diary card.
Change in OFF time | 18 months following transplantation
  Change in OFF time is measured using a Parkinson's disease patient diary card.
Change in baseline Levodopa Equivalent Daily Dose | 18 months following transplantation
  Change in Levodopa Equivalent Daily Dose (LEDD) which measures Parkinson's medications.
Change in Unified Dyskinesia Rating Scale | 18 months following transplantation
  The Unified Dyskinesia Rating Scale evaluates dyskinesia in patients with Parkinson's disease (range 0-104). A lower score indicates less dyskinesia.
Change in UPDRS Part II | 18 months following transplantation
  Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (UPDRS) Part II, which assesses the motor aspects of experiences of daily living in the week prior to the visit. Score range: 0-52. A lower score is associated with less disability.
Change in MoCA | 18 months following transplantation
  Change in Montreal Cognitive Assessment (MoCA), which measures various aspects of cognitive function. Score range 0-30. A higher score is associated with better cognitive function.
Change in DaTscan | Baseline to 18 months following transplantation
  DaTscan (SPECT neuroimaging for dopamine transporter, DAT) imaging is performed to assess changes in dopamine neuron function in the putamen (the transplanted area of the brain).

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osborn TM, Hallett PJ, Schumacher JM, Isacson O. Advantages and Recent Developments of Autologous Cell Therapy for Parkinson's Disease Patients. Front Cell Neurosci. 2020 Apr 3;14:58. doi: 10.3389/fncel.2020.00058. eCollection 2020. PMID 32317934
- [Background] Hallett PJ, Deleidi M, Astradsson A, Smith GA, Cooper O, Osborn TM, Sundberg M, Moore MA, Perez-Torres E, Brownell AL, Schumacher JM, Spealman RD, Isacson O. Successful function of autologous iPSC-derived dopamine neurons following transplantation in a non-human primate model of Parkinson's disease. Cell Stem Cell. 2015 Mar 5;16(3):269-74. doi: 10.1016/j.stem.2015.01.018. Epub 2015 Feb 26. PMID 25732245
- [Background] Hallett PJ, Cooper O, Sadi D, Robertson H, Mendez I, Isacson O. Long-term health of dopaminergic neuron transplants in Parkinson's disease patients. Cell Rep. 2014 Jun 26;7(6):1755-61. doi: 10.1016/j.celrep.2014.05.027. Epub 2014 Jun 6. PMID 24910427
- [Background] Cooper O, Hallett P, Isacson O. Using stem cells and iPS cells to discover new treatments for Parkinson's disease. Parkinsonism Relat Disord. 2012 Jan;18 Suppl 1(0 1):S14-6. doi: 10.1016/S1353-8020(11)70007-4. PMID 22166414
- [Background] Hargus G, Cooper O, Deleidi M, Levy A, Lee K, Marlow E, Yow A, Soldner F, Hockemeyer D, Hallett PJ, Osborn T, Jaenisch R, Isacson O. Differentiated Parkinson patient-derived induced pluripotent stem cells grow in the adult rodent brain and reduce motor asymmetry in Parkinsonian rats. Proc Natl Acad Sci U S A. 2010 Sep 7;107(36):15921-6. doi: 10.1073/pnas.1010209107. Epub 2010 Aug 23. PMID 20798034
- [Background] Cooper O, Astradsson A, Hallett P, Robertson H, Mendez I, Isacson O. Lack of functional relevance of isolated cell damage in transplants of Parkinson's disease patients. J Neurol. 2009 Aug;256 Suppl 3:310-6. doi: 10.1007/s00415-009-5242-z. PMID 19711122
- [Background] Mendez I, Vinuela A, Astradsson A, Mukhida K, Hallett P, Robertson H, Tierney T, Holness R, Dagher A, Trojanowski JQ, Isacson O. Dopamine neurons implanted into people with Parkinson's disease survive without pathology for 14 years. Nat Med. 2008 May;14(5):507-9. doi: 10.1038/nm1752. Epub 2008 Apr 6. PMID 18391961
- [Background] Fink JS, Schumacher JM, Ellias SL, Palmer EP, Saint-Hilaire M, Shannon K, Penn R, Starr P, VanHorne C, Kott HS, Dempsey PK, Fischman AJ, Raineri R, Manhart C, Dinsmore J, Isacson O. Porcine xenografts in Parkinson's disease and Huntington's disease patients: preliminary results. Cell Transplant. 2000 Mar-Apr;9(2):273-8. doi: 10.1177/096368970000900212. PMID 10811399
- [Background] Schumacher JM, Ellias SA, Palmer EP, Kott HS, Dinsmore J, Dempsey PK, Fischman AJ, Thomas C, Feldman RG, Kassissieh S, Raineri R, Manhart C, Penney D, Fink JS, Isacson O. Transplantation of embryonic porcine mesencephalic tissue in patients with PD. Neurology. 2000 Mar 14;54(5):1042-50. doi: 10.1212/wnl.54.5.1042. PMID 10720272
- [Background] Mendez I, Sanchez-Pernaute R, Cooper O, Vinuela A, Ferrari D, Bjorklund L, Dagher A, Isacson O. Cell type analysis of functional fetal dopamine cell suspension transplants in the striatum and substantia nigra of patients with Parkinson's disease. Brain. 2005 Jul;128(Pt 7):1498-510. doi: 10.1093/brain/awh510. Epub 2005 May 4. PMID 15872020
- [Background] Wernig M, Zhao JP, Pruszak J, Hedlund E, Fu D, Soldner F, Broccoli V, Constantine-Paton M, Isacson O, Jaenisch R. Neurons derived from reprogrammed fibroblasts functionally integrate into the fetal brain and improve symptoms of rats with Parkinson's disease. Proc Natl Acad Sci U S A. 2008 Apr 15;105(15):5856-61. doi: 10.1073/pnas.0801677105. Epub 2008 Apr 7. PMID 18391196
- [Background] Cooper O, Hargus G, Deleidi M, Blak A, Osborn T, Marlow E, Lee K, Levy A, Perez-Torres E, Yow A, Isacson O. Differentiation of human ES and Parkinson's disease iPS cells into ventral midbrain dopaminergic neurons requires a high activity form of SHH, FGF8a and specific regionalization by retinoic acid. Mol Cell Neurosci. 2010 Nov;45(3):258-66. doi: 10.1016/j.mcn.2010.06.017. Epub 2010 Jul 24. PMID 20603216